CLINICAL TRIAL: NCT01953991
Title: A Pilot Study Investigating Oral Health Related Quality of Life Improvements in Removable Partial Denture Treatments for the Replacement of Missing Teeth
Brief Title: OHQoL With Removable Partial Dentures; a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); Juvora Dental Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STH18134
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Missing Teeth; Partial Edentulism
MeSH Terms: conditions — Anodontia | interventions — Dentures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cobalt chrome dentures (Active Comparator): Cobalt chrome dentures are used as part of standard care for patients
  Interventions: Device: Dentures
- PEEK dentures (Active Comparator): PEEK dentures will be used as a comparator denture for patients
  Interventions: Device: Dentures

INTERVENTIONS:
Device: Dentures — Removable prosthesis to replace missing teeth
  Other Names: Juvora PEEK frameworks

SUMMARY:
Removable false teeth (called removable partial dentures (RPDs)) are commonly made for people with missing teeth.

RPDs are made out of a framework and the replacement teeth/gum. The framework sits on the teeth and the gums and can be made out of different materials, metal or non-metal, with different properties. The plastic teeth and gum sit on the framework.

A common framework material is cobalt chromium, a rigid, non-precious metal alloy. Other framework materials include titanium and non-metal materials such as medical grade polyetheretherketone (PEEK).

A review of the literature shows that no research has been reported investigating how different RPD framework materials impact on a person's oral health related quality of life (OHQoL). The sensation that different frameworks have in the mouth can be quite varied between people, and it would be relevant to be able to tell patients which type of framework is better tolerated based on research evidence.

We hope to conduct an un-blinded randomised crossover pilot trial investigating the difference in patient preference and oral health related quality of life measured by patient centred outcomes in a group of patients due to receive tooth supported removable partial dentures at the Charles Clifford Dental Hospital.

ELIGIBILITY:
Inclusion Criteria:

Adults from age 18 upwards:

* with the absence of 3 or more teeth, excluding third molars, per jaw arch,
* with or without previous denture wearing experience, and
* with a stable oral health in terms of absence of disease activity affecting the periodontium, dental hard tissues (caries), pulp and the structural/aesthetic integrity of restored teeth.

Exclusion Criteria:

* Patients requiring extensive treatment prior to the provision of a removable partial denture.
* Patients with active primary disease; caries, periodontal disease or symptoms of pulpal or apical pathology to the remaining teeth.
* Patients with irreversibly compromised structural/aesthetic integrity of restored teeth that cannot be restored as part of the provision of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-05; Primary Completion 2017-01-11 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Patient preference for type of denture | 6 weeks

SECONDARY OUTCOMES:
General quality of life | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Ali, BChD, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Charles Clifford Dental Hospital, Sheffield, United Kingdom